CLINICAL TRIAL: NCT03148119
Title: Phase IB Study of QRH-882260 Heptapeptide Application in the Colon
Brief Title: Study of QRH-882260 Heptapeptide Application in the Colon
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It was decided to use the QRH for a new study.
Sponsor: Danielle Kim Turgeon (Other)
Responsible Party: Sponsor-Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00122077
Record Dates: First submitted 2017-04-12; First posted 2017-05-10 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Colon Cancer Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Topical QRH Heptapeptide Administration (Experimental)
  Interventions: Drug: QRH-882260 Heptapeptide; Device: Scanning Fiber Endoscope

INTERVENTIONS:
Drug: QRH-882260 Heptapeptide — topical spray; fluorescently-labeled peptide composed of a 7-amino acid sequence [Gln-Arg-His-Lys-Pro-Arg-Glu] attached via a 5 amino acid linker [Gly-Gly-Gly-Ser-Lys] to a near-infrared fluorophore, Cy5. The complete peptide sequence is written as: Gln-Arg-His-Lys-Pro-Arg-Glu-Gly-Gly-Gly-Ser-Lys(Cy5)-NH2, and is abbreviated as: QRHKPRE-GGGSK-(Cy5)-NH2.
  Other Names: QRH
Device: Scanning Fiber Endoscope — Endoscope used for providing the light via laser to image the area of interest in the colon after the QRH has been sprayed and rinsed.

SUMMARY:
A Phase 1B study of the efficacy of a topically-administered 7-amino acid peptide labeled with a near-infrared fluorophore Cy5 for detecting neoplastic areas of the colon is proposed. The study will test the efficacy of administering this agent (QRH-882260 Heptapeptide) to human subjects undergoing clinically-indicated colonoscopy for endoscopic resection of known colonic adenomas or for surveillance biopsies of known dysplasia in the setting of irritable bowel disease (IBD). Up to 120 evaluable subjects will be enrolled.

Subjects will be recruited around scheduled standard of care procedures. The endoscopists performing the procedures are all endoscopists credentialed at the University of Michigan to do these procedures. Urine for dipstick pregnancy testing (if applicable) will be collected before the procedure, along with medical information. Vital signs are routinely monitored throughout the clinical procedure and are available in the electronic medical record. The endoscopy will proceed per the University of Michigan Health System (UMHS) standard of care. The endoscopist performing the clinical procedure will evaluate the potential risk (if any) for the subject to continue with the procedure or study. Five mL of the reconstituted QRH-882260 Heptapeptide (~100 μM) will be sprayed onto the site of interest through a catheter in the endoscope. Five minutes after QRH-882260 Heptapeptide application, the unbound peptide will be washed off using the endogator irrigator and the residual liquid will be suctioned. Pictures with white-light and fluorescence will be taken with the scanning fiber based molecular imaging endoscopic probe inserted via the instrument channel of the standard endoscope before the QRH-882260 Heptapeptide application, immediately after application and then again after the QRH-882260 Heptapeptide will be washed off. The area of interest identified will be resected/biopsied per discretion of the endoscopist per clinical care. All specimens taken are for clinical care only (not research use) and will be sent for routine histology per UMHS standard of care.

ELIGIBILITY:
Inclusion Criteria:

Subject meets at least one of the following criteria:

* At increased risk for colorectal cancer (CRC) and colonic polyps
* Known colonic adenomas scheduled for colonic resection
* Scheduled for outpatient colonoscopy for follow up surveillance of IBD with known dysplasia or who are at high risk for high grade dysplasia
* Subject is scheduled for outpatient colonoscopy in the Medical Procedures Unit at UMHS
* Subject is medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities) Standard practice guidelines for safely proceeding with the procedure will be sufficient for the study
* Age 18 to 100 years
* Willing and able to sign informed consent

Exclusion Criteria:

Subjects with known allergy or negative reaction to Cy5 (a near-infrared fluorophore) or derivatives

* Subjects on active chemotherapy or radiation treatment
* Pregnant or trying to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of QRH-882260 Heptapeptide administration-related adverse events | 1 year
  Continued monitoring of safety in subjects as measured by the number of Adverse Event (AE) assessments, severity (grade), and relationship to the study drug (any that could be related).

SECONDARY OUTCOMES:
Efficacy of QRH-882260 Heptapeptide administration for detection of polypoid and non-polypoid colonic neoplasia | 1 year
  The test product efficacy will be assessed by evaluating the fluorescence intensified measured from suspicious regions of colonic mucosa where the fluorescently-labeled peptide (QRH-882260) is administered. Measurement of peptide binding will be evaluated by the fluorescence intensity measured from the suspicious (target) region and normal tissues (background) to produce a target-to-background ratio.

OTHER OUTCOMES:
Efficacy of QRH-882260 Heptapeptide administration for detection of dysplasia in the setting of IBD | 1 year
  The test product efficacy will be assessed by evaluating the fluorescence intensified measured from suspicious regions of colonic mucosa where the fluorescently-labeled peptide (QRH-882260) is administered. Measurement of peptide binding will be evaluated by the fluorescence intensity measured from the suspicious (target) region and normal tissues (background) to produce a target-to-background ratio.

CONTACTS AND LOCATIONS:
Overall Officials: D K Turgeon, MD, Study Director — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No